CLINICAL TRIAL: NCT02249585
Title: Effects of Neuromuscular Blockade Level and Intra-abdominal Pressure on Surgical Conditions and Cardiopulmonary Responses During Laparoscopic Colon Surgery With the Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kook Hyun Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1405-010-576
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Cardiac Index
MeSH Terms: interventions — Lower Body Negative Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- CS (Experimental): Patients who receive laparoscopic colon surgery under Trendelenberg position with conventional neuromuscular blockade and standard abdominal pressure.
  Interventions: Device: Standard abdominal pressure; Drug: Conventional neuromuscular blockade
- DS (Experimental): Patients who receive laparoscopic colon surgery under Trendelenberg position with deep neuromuscular blockade and standard abdominal pressure.
  Interventions: Device: Standard abdominal pressure; Drug: Deep neuromuscular blockade
- DL (Experimental): Patients who receive laparoscopic colon surgery under Trendelenberg position with deep neuromuscular blockade and low abdominal pressure.
  Interventions: Device: Low abdominal pressure; Drug: Deep neuromuscular blockade

INTERVENTIONS:
Device: Standard abdominal pressure — Abdominal pressure maintained 12mmHg throughout laparoscopic colon surgery
  Arms: CS; DS
Device: Low abdominal pressure — Abdominal pressure maintained 8mmHg throughout laparoscopic colon surgery
  Other Names: Abdominal pressure
  Arms: DL
Drug: Conventional neuromuscular blockade — Anesthesia induction with rocuronium 0.4mg/kg and maintenance with rocuronium 0.15mg/kg to maintain TOF 1-2 twitch
  Arms: CS
Drug: Deep neuromuscular blockade — Anesthesia induction with rocuronium 0.8mg/kg → maintenance with rocuronium 0.3mg/kg to maintain PTC 1-2 twitch
  Arms: DL; DS

SUMMARY:
The purpose of this study is to find out the effect of low abdominal pressure vs. standard abdominal pressure on the cardiac and respiratory function of the patients undergoing laparoscopic colon surgery in Trendelenberg position. It was also designed to evaluate the effect of the degree of neuromuscular blockade on the surgical condition of the patients undergoing laparoscopic colon surgery in Trendelenberg position.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic colon surgery under Trendelenberg position

Exclusion Criteria:

* ASA classification IV
* Unable to make a written, informed consent
* Allergic to neuromuscular blocking agents, anesthetics, opioids
* Patients with neuromuscular disease
* Hepatic failure
* Renal failure
* History of malignant hyperthermia
* Morbid obesity with BMI>35 kg/m2
* Patients enrolled in another clinical trials

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- CS(Conventional Block With Standard Pressure): Patients who receive laparoscopic colon surgery under Trendelenberg position with conventional neuromuscular blockade and standard abdominal pressure.
  Standard abdominal pressure: Abdominal pressure maintained 12mmHg throughout laparoscopic colon surgery
  Conventional neuromuscular blockade: Anesthesia induction with rocuronium 0.4mg/kg and maintenance with rocuronium 0.15mg/kg to maintain TOF 1-2 twitch
- DS(Deep Block With Standard Pressure): Patients who receive laparoscopic colon surgery under Trendelenberg position with deep neuromuscular blockade and standard abdominal pressure.
  Standard abdominal pressure: Abdominal pressure maintained 12mmHg throughout laparoscopic colon surgery
  Deep neuromuscular blockade: Anesthesia induction with rocuronium 0.8mg/kg → maintenance with rocuronium 0.3mg/kg to maintain PTC 1-2 twitch
- DL(Deep Block With Low Pressure): Patients who receive laparoscopic colon surgery under Trendelenberg position with deep neuromuscular blockade and low abdominal pressure.
  Low abdominal pressure: Abdominal pressure maintained 8mmHg throughout laparoscopic colon surgery
  Deep neuromuscular blockade: Anesthesia induction with rocuronium 0.8mg/kg → maintenance with rocuronium 0.3mg/kg to maintain PTC 1-2 twitch
Period: Overall Study
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Started | 43 | 44 | 44
Completed | 43 | 44 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure) | Total
Number analyzed (Participants) | 43 | 44 | 44 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (12) | 64 (11) | 62 (11) | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 28 | 80
  Male | 18 | 17 | 16 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 43 | 44 | 44 | 131

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Index
Description: Cardiac index 30 min after onset of laparoscopy. The cardiac index was measured with an arterial waveform analysis system (FloTrac/EV1000, version 4.0; Edwards Life Sciences, Irvine, CA, USA) from the radial artery.
Time Frame: 30 min after onset of laparoscopy
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Number analyzed (Participants) | 43 | 44 | 44
L/min/m^2 | 2.6 (1.0) | 2.7 (0.9) | 2.7 (0.7)

2. Secondary Outcome: Mean Arterial Blood Pressure (MBP)
Description: Mean arterial blood pressure measured during laparoscopic surgery. The mean arterial blood pressure was measured with an arterial waveform analysis system (FloTrac/EV1000, version 4.0; Edwards Life Sciences, Irvine, CA, USA) from the radial artery.
Time Frame: 1, 30, 60, 90, and 120 minutes after onset of laparoscopy
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Number analyzed (Participants) | 43 | 44 | 44
mmHg
  MBP 1 min after onset of laparoscopy | 88 (13) | 92 (12) | 90 (13)
  MBP 30 min after onset of laparoscopy | 89 (10) | 92 (14) | 91 (12)
  MBP 60 min after onset of laparoscopy | 88 (11) | 90 (14) | 89 (12)
  MBP 90 min after onset of laparoscopy | 87 (11) | 89 (10) | 88 (11)
  MBP 120 min after onset of laparoscopy | 87 (13) | 90 (10) | 88 (13)

3. Secondary Outcome: Stroke Volume Index (SVI)
Description: Stroke volume index during the surgery. The stroke volume index was measured with an arterial waveform analysis system (FloTrac/EV1000, version 4.0; Edwards Life Sciences, Irvine, CA, USA) from the radial artery.
Time Frame: 1, 30, 60, 90, 120 min after onset of laparoscopy
Measure: Mean (Standard Deviation); unit: mL/beat/m^2
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Number analyzed (Participants) | 43 | 44 | 44
mL/beat/m^2
  SVI 1 min after onset of laparoscopy | 37 (9) | 41 (12) | 38 (10)
  SVI 30 min after onset of laparoscopy | 38 (10) | 42 (12) | 40 (11)
  SVI 60 min after onset of laparoscopy | 39 (12) | 42 (12) | 40 (11)
  SVI 90 min after onset of laparoscopy | 38 (9) | 41 (11) | 39 (10)
  SVI 120 min after onset of laparoscopy | 38 (9) | 40 (12) | 39 (9)

4. Secondary Outcome: PaO2
Description: PaO2 measured during laparoscopic surgery. The PaO2 (arterial partial pressure of oxygen) was measured with the blood gas analyzer (GEM Premier 3000, Model 5700; Instrumentation Laboratory, Lexington, MA, USA).
Time Frame: 1, 30, 60, 90, and 120 minutes after onset of laparoscopy
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Number analyzed (Participants) | 43 | 44 | 44
kPa
  PaO2 1 min after onset of laparoscopy | 25 (7) | 26 (7) | 27 (7)
  PaO2 30 min after onset of laparoscopy | 25 (7) | 26 (6) | 27 (7)
  PaO2 60 min after onset of laparoscopy | 25 (6) | 26 (7) | 26 (7)
  PaO2 90 min after onset of laparoscopy | 27 (6) | 28 (5) | 25 (6)
  PaO2 120 min after onset of laparoscopy | 27 (6) | 28 (5) | 25 (7)

5. Secondary Outcome: Pulmonary Compliance
Description: Pulmonary compliance during laparoscopic surgery. The pulmonary compliance was calculated from the plateau and peak inspiratory pressures, positive end-expiratory pressure, and tidal volume measured with an anesthetic machine (Primus; Dräger, Lübeck, Germany).
Time Frame: 1, 30, 60, 90, and 120 minutes after onset of laparoscopy
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Number analyzed (Participants) | 43 | 44 | 44
mL/cmH2O
  Compliance 1 min after onset of laparoscop | 29 (7) | 29 (9) | 34 (8)
  Compliance 30 min after onset of laparoscop | 24 (6) | 25 (5) | 28 (5)
  Compliance 60 min after onset of laparoscop | 25 (6) | 25 (6) | 29 (8)
  Compliance 90 min after onset of laparoscop | 26 (7) | 25 (8) | 28 (7)
  Compliance 120 min after onset of laparoscop | 28 (7) | 28 (6) | 30 (8)

6. Secondary Outcome: Surgical Rating Scale
Description: The surgical rating scale was assessed by the surgeon and graded as a five-point scale: optimal, good, acceptable, poor, and extremely poor conditions.
Time Frame: 1 min after laparoscopic procedure
Measure: Count of Participants; unit: Participants
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Number analyzed (Participants) | 43 | 44 | 44
Participants
  Optimal | 33 | 37 | 20
  Good | 3 | 7 | 6
  Acceptable | 7 | 0 | 10
  Poor | 0 | 0 | 4
  Extremely poor | 0 | 0 | 4

ADVERSE EVENTS:
Arm/Group | CS(Conventional Block With Standard Pressure) | DS(Deep Block With Standard Pressure) | DL(Deep Block With Low Pressure)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/43 | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No